CLINICAL TRIAL: NCT00025454
Title: Phase I Trial of R115777 (NSA 702818) in Advanced Malignant Solid Tumors
Brief Title: R115777 in Treating Patients With Advanced Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: City of Hope Medical Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Purpose: Treatment
Other Study IDs: CDR0000068963; U01CA062505 (NIH); P30CA033572 (NIH); CHNMC-PHI-33; NCI-4751
Record Dates: First submitted 2001-10-11; First posted 2003-01-27 (Estimated); Last update posted 2010-02-08 (Estimated); Status verified 2010-02

CONDITIONS: Unspecified Adult Solid Tumor, Protocol Specific
Keywords: unspecified adult solid tumor, protocol specific
MeSH Terms: interventions — tipifarnib

INTERVENTIONS:
Drug: tipifarnib

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die.

PURPOSE: Phase I trial to study the effectiveness of R115777 in treating patients who have advanced solid tumors.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the maximum tolerated dose of R115777 in patients with advanced malignant solid tumors.
* Assess the toxicity of this drug in these patients.
* Determine, preliminarily, the efficacy of this drug in these patients.
* Determine the potential predictors of response in patients treated with drug.

OUTLINE: This is a multicenter, dose-escalation study.

Patients receive oral R115777 twice daily on weeks 1 and 3. Treatment repeats every 28 days in the absence of disease progression or unacceptable toxicity.

Cohorts of 3-6 patients receive escalating doses of R115777 until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which at least 2 of 3 or 2 of 6 patients experience dose-limiting toxicity.

PROJECTED ACCRUAL: A minimum of 20 patients will be accrued for this study within 12 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed malignant tumors deemed to be incurable or refractory to therapy

  * Advanced, recurrent, or metastatic disease
* Previously treated with at least 1 chemotherapy regimen
* Brain metastases allowed if asymptomatic and controlled (e.g., after prior surgical resection or radiotherapy/radiosurgery) and not on steroids or anticonvulsants

PATIENT CHARACTERISTICS:

Age:

* 18 and over

Performance status:

* Karnofsky 60-100%

Life expectancy:

* Not specified

Hematopoietic:

* WBC at least 3,500/mm3
* Absolute granulocyte count at least 1,500/mm3
* Platelet count at least 75,000/mm3

Hepatic:

* Bilirubin no greater than 2.5 times upper limit of normal (ULN)
* SGOT no greater than 2.5 times ULN

Renal:

* Creatinine clearance at least 60 mL/min OR
* Creatinine no greater than 1.6 mg/dL

Other:

* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception during and for 3 months after study

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* No concurrent biologic therapy

Chemotherapy:

* See Disease Characteristics
* At least 4 weeks since prior chemotherapy (6 weeks for mitomycin or nitrosourea)

Endocrine therapy:

* See Disease Characteristics
* No concurrent hormonal therapy

Radiotherapy:

* See Disease Characteristics
* At least 4 weeks since prior radiotherapy and recovered
* No prior radiotherapy to a field containing a measurable target lesion unless there is evidence of progression or a new lesion is present
* No concurrent radiotherapy to measurable lesions

Surgery:

* See Disease Characteristics
* At least 3 weeks since prior major surgery and recovered

Other:

* At least 2 weeks since prior proton pump inhibitors (e.g., omeprazole)
* Concurrent H2 blockers (e.g., cimetidine or related drugs) or antacids are allowed if there is an interval of at least 2 hours between H2 blocker/antacid intake and R115777 dosing

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2001-08; Primary Completion 2008-07 (Actual); Study Completion 2008-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Primo N. Lara, MD, Study Chair — University of California, Davis
Locations (4):
- United States (4):
  - City of Hope Comprehensive Cancer Center, Duarte, California
  - USC/Norris Comprehensive Cancer Center and Hospital, Los Angeles, California
  - City of Hope Medical Group, Pasadena, California
  - University of California Davis Cancer Center, Sacramento, California

REFERENCES:
- [Result] Lara PN Jr, Law LY, Wright JJ, Frankel P, Twardowski P, Lenz HJ, Lau DH, Kawaguchi T, Gumerlock PH, Doroshow JH, Gandara DR. Intermittent dosing of the farnesyl transferase inhibitor tipifarnib (R115777) in advanced malignant solid tumors: a phase I California Cancer Consortium Trial. Anticancer Drugs. 2005 Mar;16(3):317-21. doi: 10.1097/00001813-200503000-00011. PMID 15711184